CLINICAL TRIAL: NCT04472871
Title: Feasibility and Prognostic Role of Percutaneous Left Atrial Appendage Closure in Patients With Heart Failure and Atrial Fibrillation at High Risk for Cerebrovascular Events
Brief Title: Feasibility and Prognosis of Left Atrial Appendage Closure in Patients With Heart Failure and Atrial Fibrillation
Acronym: LAAOHF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osman Abdelhamead, Principal Investigator, Assiut University
Other Study IDs: LAA closure in heart failure
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Device Occlusion
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- patients with atrial fibrillation and heart failure: Patients with cardiac function ejection fraction less than 35% and underwent Left atrial appendage closure in the period covered by the study
  Interventions: Device: Left atrial appendage closure
- patients with atrial fibrillation without heart failure: Patients with cardiac function ejection fraction more than 35% and underwent Left atrial appendage closure in the period covered by the study
  Interventions: Device: Left atrial appendage closure

INTERVENTIONS:
Device: Left atrial appendage closure — The left atrial appendage (LAA) is a small, ear-shaped sac in the muscle wall of the left atrium (top left chamber of the heart). It is unclear what function, if any, the LAA performs. In patients with heart failure and atrial fibrillation, reduced left atrial appendage (LAA) emptying velocities leads to LAA thrombus formation therefor a higher rate of stroke and embolism are observed even on oral anticoagulants. FDA approved devices for left atrial appendage closure will be used under guidance of angiography and trans-esophageal echo with highly efficient and trained personnel.

SUMMARY:
Study hypotheses is that in patients with heart failure and atrial fibrillation, reduced left atrial appendage (LAA) emptying velocities leads to LAA thrombus formation therefore a higher rate of stroke and embolism are observed even on oral anticoagulants.

Therefore The left atrial appendage closure (LAAC) procedure's benefit in patients with an impaired left ventricular ejection fraction (LVEF) has to be investigated So the study is to assess the safety and prognosis of left atrial appendage closure (LAAC) in patients with heart failure in preventing thromboembolic events, bleeding and all-cause mortality.

Patients will be divided into to groups, one group includes patients with no evidence of heart failure, and another group including patients with previous history of or with an evidence of with heart failure.

DETAILED DESCRIPTION:
Patients selection All patients underwent left atrial appendage closure in Assiut university in the period from January 2014 to December 2019 will be included.

Inclusion criteria In this retrospective cohort study, atrial fibrillation patients with previous major bleeding, bleeding predisposition or contraindications for oral anticoagulants scheduled for transcatheter left atrial appendage closure are included.

Methods In this retrospective cohort study

1. All patients with previous major bleeding or a bleeding predisposition scheduled for transcatheter LAAC in Assiut university in the period from January 2014 to December 2019 will be included.
2. All devices used in for LAAC in this period will be included (WATCHMAN, Amulet, LARIAT and Lambre)
3. CHA2DS2-VASC, CHADS, HAS-BLED scores will be calculated for all patients.
4. Patients will be divided into to groups, one group includes patients with no evidence of heart failure, and another group including patients with previous history of or with an evidence of with heart failure.
5. Heart failure will be defined as patients with left ventricular ejection fraction ≤ 35%.
6. New York Heart Association (NYHA) classification will be determined for all patient graded from I-IV.
7. Both groups will be compared regarding procedural success (Procedural success is defined as deployment and release of the left atrial appendage closure device into the LAA with peri-device leak < 5 mm), the absence of any complication related to the intervention, major and minor bleeding, all-cause mortality and efficacy of the device to prevent stroke, transient ischemic attack, systemic embolization during follow-up.
8. Device related thrombus (DRT) will be compared in both groups according to the results of transesophageal echo (TOE) 6 weeks post procedure.

Primary endpoint

- The primary endpoints of the study are procedural success (Procedural success is defined as deployment and release of the left atrial appendage closure device into the LAA with peri-device leak < 5 mm), the absence of any complication related to the intervention, bleeding, all-cause mortality and efficacy of the device to prevent stroke, transient ischemic attack, systemic embolization during follow-up in both groups of patients with heart failure and without heart failure.

ELIGIBILITY:
Inclusion Criteria:

* In this study,

  1. Atrial fibrillation patients with previous major bleeding.
  2. Atrial fibrillation patients with previous bleeding predisposition
  3. Atrial fibrillation patients with previous contraindications for oral anticoagulants scheduled for transcatheter left atrial appendage closure are included.

Exclusion Criteria:

* Patients having no data for follow up after the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent left atrial appendage closure in Assiut university in the period from January 2014 to December 2019 will be included.
  In this retrospective cohort study, atrial fibrillation patients with previous major bleeding, bleeding predisposition or contraindications for oral anticoagulants who were scheduled for transcatheter left atrial appendage closure are included
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
procedural success | 6 weeks post procedure
  procedural success (Procedural success is defined as deployment and release of the left atrial appendage closure device into the LAA with peri-device leak < 5 mm) The study will assess the rate of procedural success in both groups of the study.
the absence of any complication related to the intervention | 6 months post intervention
  Post procedural Complications including cerebrovascular stroke, bleeding and all cause mortality will be compared in both groups of the study to assess the prognosis of the procedure in these groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Osman, Ass. lect., Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Result] Holmes DR Jr, Doshi SK, Kar S, Price MJ, Sanchez JM, Sievert H, Valderrabano M, Reddy VY. Left Atrial Appendage Closure as an Alternative to Warfarin for Stroke Prevention in Atrial Fibrillation: A Patient-Level Meta-Analysis. J Am Coll Cardiol. 2015 Jun 23;65(24):2614-2623. doi: 10.1016/j.jacc.2015.04.025. PMID 26088300
- [Result] Saw J. Long-Term Results With Left Atrial Appendage Closure: Watching the Watchman. J Am Coll Cardiol. 2017 Dec 19;70(24):2976-2978. doi: 10.1016/j.jacc.2017.10.056. Epub 2017 Nov 2. No abstract available. PMID 29104013
- [Result] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Result] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Result] Ellis CR, Kanagasundram AN. Atrial Fibrillation in Heart Failure: Left Atrial Appendage Management. Cardiol Clin. 2019 May;37(2):241-249. doi: 10.1016/j.ccl.2019.01.009. Epub 2019 Feb 13. PMID 30926025